CLINICAL TRIAL: NCT04994782
Title: GAMification to Encourage End-Of-Life Discussions Between Implantable Cardioverter Defibrillator Recipients and Family Members
Brief Title: GAMification to Encourage End-Of-Life Discussions Between ICD Patients and Caregivers
Acronym: GAME-EOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Debra Moser (Other)
Collaborators: University of Kentucky CCTS (Unknown)
Responsible Party: Sponsor-Investigator, Debra Moser, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 61699
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Implantable Defibrillator User; Terminal Illness
Keywords: End-of-life; Healthcare Communication; Advance Directives
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care recipients (No Intervention): Participant dyads in this group will receive usual care (standard clinical education materials)
- Usual care plus GAME-EOL intervention (Experimental): Participant dyads in this group will receive usual care (standard clinical education materials) plus the GAME-EOL intervention.
  Interventions: Behavioral: GAME-EOL

INTERVENTIONS:
Behavioral: GAME-EOL — The GAME-EOL involves Hello game booklets as well as meetings with an interventionist. Players (ICD recipient and their family member or friend dyad) take turns asking the questions in their booklet and providing their answers to the question. The gameplay continues until all questions are answered or the dyad wishes to stop. Following the completion of the game play, participants will be offered the opportunity to complete advance directives using the conversation guide and advance directive form included in the conversation guide that accompanies the questionnaire booklet.
  Arms: Usual care plus GAME-EOL intervention

SUMMARY:
The purpose of this study is to determine the feasibility and efficacy of the GAMification to Encourage End-Of-Life (GAME-EOL) intervention, which uses the Hello Game program to encourage and facilitate quality end-of-life (EOL) discussions between implantable cardioverter defibrillators (ICD) recipients and family members of ICD recipients.

DETAILED DESCRIPTION:
Implantable cardioverter defibrillators (ICD)s are first-line treatment for the primary and secondary prevention of sudden cardiac arrest in populations with a history of, or at high risk for, lethal arrhythmias. Despite the relatively short survival expectancy following device implantation, many ICD recipients do not participate in advance care planning and either have no advance directives or advance directives that do not address end-of-life (EOL) decisions related to ICDs. The prevalence of ICD recipients with general advance directives ranges from 10-30%. Of these advance directives, only 2% have language related to the ICD specifically, leaving hundreds of thousands of ICD recipients at risk of unnecessary and painful shocks. Approximately 30% of ICD recipients will receive a shock in the active dying phase of a terminal illness, from which resuscitation was not intended.

Communication among family members is integral to EOL decision-making. Appropriate quality discussions can create concordance of perceptions and well thought out advance care plans for EOL that are congruent with the values and beliefs of the chronically ill and family members. The Hello Game (commonpractice.com) was created to encourage conversations among families about EOL choices. The gameplay presents a series of questions that include practical and philosophical question prompts. These questions range from 1) What kind of music would you like to be listening to on your last day alive? to 2) Who should your health care surrogate seek advice from if they need to make a decision about your care? Participation in the game has been found to improve advance care planning behaviors.

The purpose of this pilot study is to determine the feasibility and efficacy of the GAME-EOL intervention, which uses the Hello Game to encourage and facilitate quality EOL discussions between ICD recipients and family members.

Aim 1: To determine feasibility of the GAME-EOL intervention to facilitate EOL conversations between ICD recipients and family members.

Aim 2: To provide preliminary estimates of the efficacy of the GAME-EOL intervention on: (2.1) Completion of advance directives (2.2) Completion of device specific advance directives (2.3) Discussion of EOL choices between ICD recipients and family members

Aim 3: To examine efficacy of GAME-EOL on improving the concordance of EOL perceptions and advance care planning between ICD recipients and family members.

ELIGIBILITY:
Inclusion Criteria:

* ICD recipients with a family member or friend who lives with them or provides a significant role in the healthcare decision making process
* Internet access

Exclusion Criteria:

* Age less than 18 years
* No family member or friend willing to participate with the ICD recipient
* Significant cognitive impairment
* Institutionalization (e.g., nursing home, prison)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of GAME-EOL | At study completion, up to 3 months post intervention
  The feasibility, likability, and acceptability of GAME-EOL will be assessed using a Likert style questionnaire and one open-ended question. Recruitment and retention statistics will be calculated to provide additional quantitative assessment of feasibility and acceptability.
  This questionnaire consists of 18 Likert style questions and one open-response section allowing participants to place additional comments. These questions are broken down into six categories: 1) four questions relating to the content of the education and intervention sessions, 2) four questions related to the technology used to collect data (it's feasibility and user-friendliness), 3) three questions related to the intervention itself, 4) four questions related to the effectiveness of the instructional methodology, 5) three questions about the participants comfort level throughout the study, and 6) one section for additional comments
Completion of Advance Directives | 8 weeks post intervention
  The prevalence of completed general and device specific advance directives will be compared to reports in the literature to determine effectiveness. Medical records will be reviewed eight weeks following completion of data collection to determine if the advance directives were communicated to the healthcare provider and placed in the participants' electronic medical record. Additionally, 8 weeks following study completion, the participants will be contacted for a self-report of conversations with healthcare providers and family.
Change in concordance of end of life (EOL) Attitudes | Baseline, post intervention
  The Preferences for Care Near the End-of-Life instrument will be used to determine congruence of EOL attitudes between ICD recipient and family member. This 32-item questionnaire uses a 5-point Likert scale to identify attitudes toward EOL care with questions such as "I do not want CPR" and "I want my family to make all of my decisions". The instrument will be completed by the ICD recipient and an adapted version with the stem of the question changed from "I" to "my family member" will be completed by family members. Completed instruments will be compared to determine the convergence of attitudes and clarity of communication that occurred during the intervention. This instrument has been found to be valid and reliable in multiple populations. This instrument will be completed by both patients and family members.
Change in experience of end of life issues | Baseline, post intervention
  This 10 item subscale of the ICD End-of-Life Questionnaire assesses the experiences of end of life issues using a 5-point Likert scale ranging from 'Not at all' to 'Very much so'. These questions center around a participant's or Caregiver's worries about the ICD device in every-day and EOL contexts. These questions will be asked at the initial Baseline assessment and then again after the education/intervention. The differences in experiences and worries will be assessed. A higher score (the 'Very much so' option) relates to higher levels of worry and anxiety about their device.
  This instrument will be completed by both patients and family members.
Change in attitudes about discussions and actions related to end of life | Baseline, post intervention
  This 18 item subscale of the ICD End-of-Life Questionnaire assesses the attitudes about discussions and actions related to end of life, which break down into two categories. For the first 10 questions, patients can select either 'Agree' or Disagree'. These assess the attitudes a participant has about discussing, with a healthcare professional, the issue of turning off the ICD in the event they are experiencing painful shocks. The remaining 8 questions are intended to assess their attitudes toward the ICD itself in the context of deteriorated health. Participants have the choice of selecting 'Yes', 'No', and 'Can't take a stand'. We will also qualitatively analyze the recorded interventions to detect any change of attitudes about EOL topics.
  This instrument will be completed by both patients and family members.
Knowledge about the ICD in relation to end of life (EOL). | Baseline, post intervention
  This 11 item subscale of the ICD End-of-Life Questionnaire assesses the knowledge about the ICD in relation to EOL. It contains 11 items divided into ethical aspects, function of the ICD, and practical consequences, and has been shown to be valid and reliable in the ICD recipient and caregiver populations. This will be administered before and after the intervention so that we may see the effects of the intervention and education on the patient's/caregiver's understanding of their device. For each question, participants can either select 'True', 'False', or 'Don't know'.
  This instrument will be completed by both patients and family members.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Moser, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Kramer DB, Kennedy KF, Noseworthy PA, Buxton AE, Josephson ME, Normand SL, Spertus JA, Zimetbaum PJ, Reynolds MR, Mitchell SL. Characteristics and outcomes of patients receiving new and replacement implantable cardioverter-defibrillators: results from the NCDR. Circ Cardiovasc Qual Outcomes. 2013 Jul;6(4):488-97. doi: 10.1161/CIRCOUTCOMES.111.000054. Epub 2013 Jun 11. PMID 23759471
- [Background] Sherazi S, McNitt S, Aktas MK, Polonsky B, Shah AH, Moss AJ, Daubert JP, Zareba W. End-of-life care in patients with implantable cardioverter defibrillators: a MADIT-II substudy. Pacing Clin Electrophysiol. 2013 Oct;36(10):1273-9. doi: 10.1111/pace.12188. Epub 2013 Jun 3. PMID 23731284
- [Background] Tajouri TH, Ottenberg AL, Hayes DL, Mueller PS. The use of advance directives among patients with implantable cardioverter defibrillators. Pacing Clin Electrophysiol. 2012 May;35(5):567-73. doi: 10.1111/j.1540-8159.2012.03359.x. Epub 2012 Mar 20. PMID 22432897
- [Background] Merchant FM, Binney Z, Patel A, Li J, Peddareddy LP, El-Chami MF, Leon AR, Quest T. Prevalence, predictors, and outcomes of advance directives in implantable cardioverter-defibrillator recipients. Heart Rhythm. 2017 Jun;14(6):830-836. doi: 10.1016/j.hrthm.2017.02.022. Epub 2017 Feb 20. PMID 28232262
- [Background] Kinch Westerdahl A, Sjoblom J, Mattiasson AC, Rosenqvist M, Frykman V. Implantable cardioverter-defibrillator therapy before death: high risk for painful shocks at end of life. Circulation. 2014 Jan 28;129(4):422-9. doi: 10.1161/CIRCULATIONAHA.113.002648. Epub 2013 Nov 15. PMID 24243857
- [Background] Westerdahl AK, Sutton R, Frykman V. Defibrillator patients should not be denied a peaceful death. Int J Cardiol. 2015 Mar 1;182:440-6. doi: 10.1016/j.ijcard.2015.01.012. Epub 2015 Jan 6. PMID 25597981
- [Background] Miller JL. Social Determinants of Health and Disparities in Outcomes Related to Cardiovascular Health inVulnerable Populations. Nursing. 2017;PhD:204.
- [Background] Scott AM, Caughlin JP. Communication nonaccommodation in family conversations about end-of-life health decisions. Health Commun. 2015;30(2):144-53. doi: 10.1080/10410236.2014.974128. PMID 25470439
- [Background] Weiner JS, Roth J. Avoiding iatrogenic harm to patient and family while discussing goals of care near the end of life. J Palliat Med. 2006 Apr;9(2):451-63. doi: 10.1089/jpm.2006.9.451. PMID 16629574
- [Background] Lautrette A, Darmon M, Megarbane B, Joly LM, Chevret S, Adrie C, Barnoud D, Bleichner G, Bruel C, Choukroun G, Curtis JR, Fieux F, Galliot R, Garrouste-Orgeas M, Georges H, Goldgran-Toledano D, Jourdain M, Loubert G, Reignier J, Saidi F, Souweine B, Vincent F, Barnes NK, Pochard F, Schlemmer B, Azoulay E. A communication strategy and brochure for relatives of patients dying in the ICU. N Engl J Med. 2007 Feb 1;356(5):469-78. doi: 10.1056/NEJMoa063446. PMID 17267907
- [Background] Detering KM, Hancock AD, Reade MC, Silvester W. The impact of advance care planning on end of life care in elderly patients: randomised controlled trial. BMJ. 2010 Mar 23;340:c1345. doi: 10.1136/bmj.c1345. PMID 20332506
- [Background] Ahrens T, Yancey V, Kollef M. Improving family communications at the end of life: implications for length of stay in the intensive care unit and resource use. Am J Crit Care. 2003 Jul;12(4):317-23; discussion 324. PMID 12882061
- [Background] Parks SM, Winter L, Santana AJ, Parker B, Diamond JJ, Rose M, Myers RE. Family factors in end-of-life decision-making: family conflict and proxy relationship. J Palliat Med. 2011 Feb;14(2):179-84. doi: 10.1089/jpm.2010.0353. Epub 2011 Jan 21. PMID 21254816
- [Background] Siminoff LA, Rose JH, Zhang A, Zyzanski SJ. Measuring discord in treatment decision-making; progress toward development of a cancer communication and decision-making assessment tool. Psychooncology. 2006 Jun;15(6):528-40. doi: 10.1002/pon.989. PMID 16206332
- [Background] The Hello Game. 2019.
- [Background] Van Scoy LJ, Reading JM, Hopkins M, Smith B, Dillon J, Green MJ, Levi BH. Community Game Day: Using an End-of-Life Conversation Game to Encourage Advance Care Planning. J Pain Symptom Manage. 2017 Nov;54(5):680-691. doi: 10.1016/j.jpainsymman.2017.07.034. Epub 2017 Jul 23. PMID 28743662
- [Background] Radhakrishnan K, Van Scoy LJ, Jillapalli R, Saxena S, Kim MT. Community-based game intervention to improve South Asian Indian Americans' engagement with advanced care planning. Ethn Health. 2019 Aug;24(6):705-723. doi: 10.1080/13557858.2017.1357068. Epub 2017 Jul 27. PMID 28748743
- [Background] Al-Khatib SM, Stevenson WG, Ackerman MJ, Bryant WJ, Callans DJ, Curtis AB, Deal BJ, Dickfeld T, Field ME, Fonarow GC, Gillis AM, Granger CB, Hammill SC, Hlatky MA, Joglar JA, Kay GN, Matlock DD, Myerburg RJ, Page RL. 2017 AHA/ACC/HRS guideline for management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Heart Rhythm. 2018 Oct;15(10):e73-e189. doi: 10.1016/j.hrthm.2017.10.036. Epub 2017 Oct 30. No abstract available. PMID 29097319
- [Background] Gadoud A, Jenkins SM, Hogg KJ. Palliative care for people with heart failure: summary of current evidence and future direction. Palliat Med. 2013 Oct;27(9):822-8. doi: 10.1177/0269216313494960. Epub 2013 Jul 9. PMID 23838375
- [Background] Rogers JG, Patel CB, Mentz RJ, Granger BB, Steinhauser KE, Fiuzat M, Adams PA, Speck A, Johnson KS, Krishnamoorthy A, Yang H, Anstrom KJ, Dodson GC, Taylor DH Jr, Kirchner JL, Mark DB, O'Connor CM, Tulsky JA. Palliative Care in Heart Failure: The PAL-HF Randomized, Controlled Clinical Trial. J Am Coll Cardiol. 2017 Jul 18;70(3):331-341. doi: 10.1016/j.jacc.2017.05.030. PMID 28705314
- [Background] Caughlin JP. Multiple Goals Theory of Personal Relationships: Conceptual Integration and Program Overview. Journal of Social and Personal Relationships. 2010;27:824-848.
- [Background] Thylen I, Wenemark M, Fluur C, Stromberg A, Bolse K, Arestedt K. Development and evaluation of the EOL-ICDQ as a measure of experiences, attitudes and knowledge in end-of-life in patients living with an implantable cardioverter defibrillator. Eur J Cardiovasc Nurs. 2014 Apr;13(2):142-51. doi: 10.1177/1474515113515563. Epub 2013 Dec 1. PMID 24298191
- [Background] Gauthier DM, Froman RD. Preferences for care near the end of life: scale development and validation. Res Nurs Health. 2001 Aug;24(4):298-306. doi: 10.1002/nur.1031. PMID 11746060
- [Background] Schirm V, Sheehan D, Zeller RA. Preferences for Care Near the End of Life: instrument validation for clinical practice. Crit Care Nurs Q. 2008 Jan-Mar;31(1):24-32. doi: 10.1097/01.CNQ.0000306393.79282.5b. PMID 18316933
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Kroenke K and Spitzer RL. The PHQ-9: A new depression diagnostic and severity measure. Psychiatric Annals. 2002;32:1-7.
- [Background] Hammash MH, Hall LA, Lennie TA, Heo S, Chung ML, Lee KS, Moser DK. Psychometrics of the PHQ-9 as a measure of depressive symptoms in patients with heart failure. Eur J Cardiovasc Nurs. 2013 Oct;12(5):446-53. doi: 10.1177/1474515112468068. Epub 2012 Dec 21. PMID 23263270
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Resnick B, Parker R. Simplified scoring and psychometrics of the revised 12-item Short-Form Health Survey. Outcomes Manag Nurs Pract. 2001 Oct-Dec;5(4):161-6. PMID 11898312
- [Background] Frizelle DJ, Lewin B, Kaye G, Moniz-Cook ED. Development of a measure of the concerns held by people with implanted cardioverter defibrillators: the ICDC. Br J Health Psychol. 2006 May;11(Pt 2):293-301. doi: 10.1348/135910705X52264. PMID 16643700
- [Background] Weiss BD, Mays MZ, Martz W, Castro KM, DeWalt DA, Pignone MP, Mockbee J, Hale FA. Quick assessment of literacy in primary care: the newest vital sign. Ann Fam Med. 2005 Nov-Dec;3(6):514-22. doi: 10.1370/afm.405. PMID 16338915
- [Background] Osborn CY, Weiss BD, Davis TC, Skripkauskas S, Rodrigue C, Bass PF, Wolf MS. Measuring adult literacy in health care: performance of the newest vital sign. Am J Health Behav. 2007 Sep-Oct;31 Suppl 1:S36-46. doi: 10.5555/ajhb.2007.31.supp.S36. PMID 17931135
- [Background] Rayens MK, Svavarsdottir EK. A new methodological approach in nursing research: an actor, partner, and interaction effect model for family outcomes. Res Nurs Health. 2003 Oct;26(5):409-19. doi: 10.1002/nur.10100. PMID 14579261
- [Background] Cohen J. Statistical power analysis for the behavioral sciences Lawrence Erlbaum Associates; 1988.